CLINICAL TRIAL: NCT03706573
Title: Managed Access Program (MAP) to Provide Alpelisib for Patients With HR+ Advanced or Metastatic Breast Cancer Resistant or Refractory to Available Treatment Options
Brief Title: Managed Access Program to Provide Alpelisib for Patients With HR+ Advanced or Metastatic Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719A0US01CM
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: HR+ Advanced or Metastatic Breast Cancer
Keywords: byl719; adult; breast cancer; HR+ advanced cancer; HR+ metastic cancer; resistant; refractory
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: alpelisib — 50 mg and 200 mg film coated tablets administered orally once daily. Starting dose is 350 mg daily. Starting dose as a combination agent with endocrine partner is 300mg daily.

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to alpelisib for eligible patients diagnosed with hormone receptor positive, advanced or metastatic breast cancer harboring a phosphatidylinositol 3-kinase (PI3K)CA mutation. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient can and will sign the Informed Consent (ICF) prior to eligibility evaluations being performed and is able to comply with treatment plan requirements
2. Patient is an adult and ≥ 18 years old at the time of informed consent
3. Patient has locally advanced or metastatic HR+ breast cancer and no comparable or satisfactory alternative therapy is available
4. PIK3CA mutation in tumor tissue or ctDNA as determined by a local laboratory
5. Patient is not:

   1. eligible for participation in any ongoing clinical trials with alpelisib, or has recently completed a clinical trial with alpelisib that has been terminated
   2. being transferred from or participating in an ongoing clinical trial, and after considering other options (e.g. trial extensions, amendments, etc.), treating physician has determined that treatment is necessary and there are no other feasible alternatives for the patient
6. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L (For patients with hematologic malignancies involving the bone marrow, platelet count > 75 x 109/L may be acceptable)
   3. Hemoglobin ≥ 9.0 g/dL
   4. INR ≤ 1.5
   5. Potassium, magnesium and calcium (corrected for albumin), within normal limits for the institution, or ≤ Grade 1 severity according to NCI-CTCAE version 4.03 if judged clinically not significant by the investigator
   6. Serum creatinine ≤ 1.5 x ULN and/or creatinine clearance > 50% LLN (Lower Limit of Normal)
   7. Total serum bilirubin < ULN (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome, (defined as presence of several episodes of unconjugated hyperbilirubinemia with normal CBC results including normal reticulocyte count and peripheral blood smear, normal liver function test results, and absence of other contributing disease processes at the time of diagnosis)
   8. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 ULN (or < 5.0 x ULN if liver metastases are present)
   9. Fasting plasma glucose (FPG) ≤ 140mg/dL or ≤ 7.7 mmol/L* or Glycosylated Hemoglobin (HbA1c)≤ 6.4% (both criteria have to be met).
7. Patient is deemed by the Treating Physician to have the initiative and means to be compliant with the treatment plan (treatment and follow-up requested by the Treating Physician)

Exclusion Criteria:

1. Patient has history of hypersensitivity to any drugs or metabolites of PI3K inhibitor.
2. Patient has not recovered to grade 1 or better (except alopecia) from side effects of any prior antineoplastic therapy
3. Patient has had major surgery within 14 days prior to starting treatment with alpelisib or has not recovered from major side effects
4. Patient is currently receiving high doses of systemic corticosteroids ≤ 2 weeks prior to starting treatment with alpelisib, or has not fully recovered from side effects of such treatment. (Note: low dose corticosteroids are permitted: single doses, topical applications, inhaled sprays, eye applications or local injections, stable low dose, for patients with CNS tumors, for at least 2 weeks prior to start of alpelisib treatment.)
5. Patient with uncontrolled diabetes mellitus.
6. Patient is being treated at start of treatment with alpelisib with any of the following drugs:

   Drugs known to be strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications (list of prohibited CYP3A4 inhibitors and inducers provided in Table 13-2 in Appendix) Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment with alpelisib is initiated. Switching to a different medication prior to starting treatment with alpelisib is allowed.
7. Patient is currently receiving warfarin or other coumarin derived anti-coagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed. Patients receiving therapies listed in Table 13-2 would not be allowed.
8. Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgment, contraindicate patient participation in the individual patient program (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
9. Patient has a known history of Steven Johnson's syndrome or toxic epidermal necrolysis
10. Patient with active HIV infection (testing not mandatory) infection
11. Patient has any of the following cardiac abnormalities:

    1. symptomatic congestive heart failure
    2. history of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
    3. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
    4. myocardial infarction ≤ 6 months prior to enrolment
    5. unstable angina pectoris
    6. serious uncontrolled cardiac arrhythmia
    7. symptomatic pericarditis
12. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of alpelisib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Hester A, Henze F, Travi C, Harbeck N, Wuerstlein R. First Experiences with Alpelisib in Clinical Routine: Case Reports from a German Breast Center. Breast Care (Basel). 2021 Apr;16(2):129-134. doi: 10.1159/000514794. Epub 2021 Mar 15. PMID 34012367